CLINICAL TRIAL: NCT01015235
Title: A Double-Blind, Randomized, Placebo- and Active-Comparator-Controlled, Single-Dose Study to Assess the Efficacy of KAI-1678 Administered by Subcutaneous Infusion for the Treatment of Postoperative Pain
Brief Title: Safety and Efficacy Study of KAI-1678 to Treat Subjects With Postoperative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KAI Pharmaceuticals (Industry)
Collaborators: Trident Clinical Research Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAI-1678-002
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Pain, Postoperative
Keywords: Ketorolac / therapeutic use; Analgesics. Non-narcotic / therapeutic use; Arthroplasty, replacement hip; Arthroplasty, replacement knee; Pain measurement / drug effect; Pain postoperative / drug therapy
MeSH Terms: conditions — Pain, Postoperative | interventions — KAI-1678; Bulk Drugs; Ketorolac Tromethamine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- A2: KAI-1678 (Active Comparator): Test Drug
  Interventions: Drug: KAI-1678
- A3: Ketorolac (Active Comparator): Active Comparator
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Placebo — Subcutaneous infusion-once over 4 hours
  Arms: Arm 1: Placebo
Drug: KAI-1678 — Subcutaneous infusion-once over 4 hours
  Other Names: Active drug
  Arms: A2: KAI-1678
Drug: Ketorolac Tromethamine — Active comparator, IV infusion, once
  Other Names: Ketorolac
  Arms: A3: Ketorolac

SUMMARY:
The purpose of this study is to determine whether KAI-1678 is effective in the treatment of postoperative pain following total hip or total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) classification 1, 2, or 3
* total hip or total knee replacement
* pain on postoperative Day 1 at least 40 mm on 0-100 mm visual analog scale (VAS)

Exclusion Criteria:

* presence of contraindications to nonsteroidal anti-inflammatory (NSAID) treatment
* recent history of angina or myocardial infarction (MI)
* clinically significant abnormality on laboratory tests or electrocardiogram (ECG)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The effect of KAI-1678 on summed pain intensity difference over 4 hours (SPID 4). | Post operative Day 1

SECONDARY OUTCOMES:
The effect of KAI-1678 on total pain relief over 4 hours (TOTPAR 4) | Post operative Day 1
The effect of KAI-1678 on pain intensity difference (PID) at 4 hours | Post-operative Day 1
The effect of KAI-1678 on total quality analgesia | Post-operative Day 1
The effect of KAI-1678 on time to meaningful pain relief | Post-operative Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Bell, MD, Study Director — KAI Pharmaceuticals
Locations (1):
- Hamilton, New Zealand